CLINICAL TRIAL: NCT01650337
Title: Randomized Trial of a Smartphone Application for Weight Loss in Primary Care
Brief Title: mFit: The Mobile Fitness Project
Acronym: mFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Brian Y. Laing, Robert Wood Johnson Clinical Scholar, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: mFit-UCLA
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Overweight; Obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smartphone Application (Experimental): Patients will be given access to a smartphone application for weight loss and instructed on how to use it.
  Interventions: Other: Smartphone Application
- Usual primary care (No Intervention)

INTERVENTIONS:
Other: Smartphone Application — Smartphone application to help monitor caloric intake and expenditure
  Arms: Smartphone Application

SUMMARY:
BACKGROUND: The nascent field of mobile health (mHealth) is expanding with impressive speed. In March 2012, experts estimated that 40,000 health related smartphone applications were on the market but little is known about the effectiveness of these programs. To our knowledge, no studies have evaluated whether weight loss can be successfully achieved through use of a smartphone application or how these applications could be used in primary care practice.

PURPOSE: To evaluate the effectiveness of a popular, free smartphone application for weight loss and calorie counting in a primary care setting.

METHODS: The first phase of this study involved a community based participatory approach to select the intervention. Patient focus groups were conducted and analyzed to explore patients' preferences regarding various text-message versus smartphone programs. The second phase of this study, described here, will be a randomized controlled trial with overweight primary care patients exposed to one of two conditions for 6 months: (1) usual care; (2) usual care plus smartphone application, which includes instructing participants on how to use the application and encouraging them to use the applications' reminders and social networking features. The primary outcome of interest is weight change at 3 and 6 months. Two-sample t-test or Wilcoxon rank sum test will be used to compare weight change between groups, as appropriate. ANCOVA models will be used to examine weight change after adjusting for covariates such as education, sex and age. Repeated measures analysis will be carried out to compare weight change between the groups using baseline, 3 month and 6 month data. In addition to an intent-to-treat analysis, the investigators will also conduct a "treatment received" analysis, adjusting for the extent of application use in both the intervention and control arms.

CONCLUSIONS: This study will demonstrate whether a smartphone application introduced in primary care settings and incorporated into the visit can produce weight loss. Study findings could inform a national discourse on the value of smartphone applications in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* primary care patient at UCLA Family Health Center or 16th Street Internal Medicine
* age 18 or older,
* English speaking,
* BMI > 25,
* interested in losing weight,
* smartphone ownership,
* valid email address.

Exclusion Criteria:

* current, planned or previous pregnancy within 6 months,
* currently using a smartphone app for dieting,
* hemodialysis,
* terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
weight loss | six months

SECONDARY OUTCOMES:
systolic blood pressure | six months

OTHER OUTCOMES:
Self-efficacy in dieting | six months
  Based on 2 questions adapted from the diabetes empowerment scale (DES)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Y Laing, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA Family Health Center, Santa Monica, California
  - UCLA Internal Medicine, Santa Monica, California

REFERENCES:
- [Derived] Laing BY, Mangione CM, Tseng CH, Leng M, Vaisberg E, Mahida M, Bholat M, Glazier E, Morisky DE, Bell DS. Effectiveness of a smartphone application for weight loss compared with usual care in overweight primary care patients: a randomized, controlled trial. Ann Intern Med. 2014 Nov 18;161(10 Suppl):S5-12. doi: 10.7326/M13-3005. PMID 25402403